CLINICAL TRIAL: NCT01166464
Title: Examining a Text Message Intervention for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Live Inspired, LLC (Industry)
Responsible Party: Principal Investigator, Beth Bock, Ph.D., Staff Psychologist, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21DA027142 (NIH)
Record Dates: First submitted 2010-07-16; First posted 2010-07-21 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Tobacco Use Disorder; Nicotine Dependence
Keywords: tobacco; smoking; text message; therapy
MeSH Terms: conditions — Tobacco Use Disorder; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text Messaging (Experimental): A text message-based intervention for smoking cessation
  Interventions: Behavioral: text messaging for smoking cessation
- Control (Placebo Comparator): Individuals in this group will receive generic (non-smoking related) text messages on the same schedule as the intervention arm. This provides a control for staff/program contact time and participant burden.
  Interventions: Behavioral: Generic text messages

INTERVENTIONS:
Behavioral: text messaging for smoking cessation — A 7-week program of daily text messages
  Arms: Text Messaging
Behavioral: Generic text messages — non-smoking related text messages will be given on the same daily schedule as matches the active intervention to establish a control for contact time.
  Arms: Control

SUMMARY:
The primary goal of this study is to use qualitative interviews and focus groups to aid us in adapting a face-to-face smoking cessation intervention for delivery through text messaging. After design is completed, the intervention will be pilot tested with a sample of young adults (ages 18-35) who smoke. Final assessments will be conducted at 7 weeks (end of treatment) and both 3 and 6 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 35
* Current daily smoker
* Has a cell phone with text messaging capability
* Uses text messaging at least once monthly
* Interested in quitting smoking
* Willing to set a quit date within the next 30 days
* Has access to a physician

Exclusion Criteria:

* Does not read and speak English with adequate comprehension
* Is currently participating in a smoking cessation program
* Concurrent drug/alcohol abuse
* Mental health issues that would interfere with study compliance

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2009-07; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence | Six months post-treatment
  7-day point prevalence abstinence will be measured at 6 months post-treatment.

SECONDARY OUTCOMES:
Usability and Acceptability of the intervention | 7 weeks (end of treatment)
  Usability and acceptability of the intervention will be assessed at the end of treatment (week 7).

CONTACTS AND LOCATIONS:
Overall Officials: Beth C Bock, PhD, Principal Investigator — The Miriam Hospital, Brown Medical School
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Bock B, Heron K, Jennings E, Morrow K, Cobb V, Magee J, Fava J, Deutsch C, Foster R. A Text Message Delivered Smoking Cessation Intervention: The Initial Trial of TXT-2-Quit: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2013 Jul 30;1(2):e17. doi: 10.2196/mhealth.2522. PMID 25098502